CLINICAL TRIAL: NCT04321603
Title: Altering Mechanisms of Frailty in Persons Living With HIV Aged 50 to 65
Acronym: ALTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 prevented us from doing this human subjects study
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Jennifer Klinedinst, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HP-00089501
Record Dates: First submitted 2020-03-19; First posted 2020-03-25 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Hiv; Frailty Syndrome
Keywords: physical activity; mitochondrial respiration; inflammation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Frailty; Motor Activity; Inflammation | interventions — Walking; Exercise

STUDY DESIGN:
Intervention Model Description: This within-subjects design will allow each subject to be utilized as their own control pre-intervention. With expectation of great inter-person variability of oxygen consumption results, this design will incorporate less error than separately recruited controls and decrease the needed sample size.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People living with HIV (Other): Subjects will act as own control between Visit one and Visit two, then will complete six weeks of walking, 30 minutes per walk, three times weekly between Visit Two and Visit Three.
  Interventions: Behavioral: Walking

INTERVENTIONS:
Behavioral: Walking — Moderately paced walking of approximately 100 steps/minute for 30 minutes three times weekly for six weeks.
  Other Names: physical activity

SUMMARY:
People living with HIV are living longer as their disease is controlled with antiretroviral medications. Yet they are experiencing frailty more often and more than ten years earlier than those without HIV. In elderly persons without HIV, frailty is associated with decreased muscle strength and chronic inflammation. Less is known about what is driving early frailty in HIV or effective prevention measures for aging adults with HIV.

It may be that having HIV infection impairs energy production by mitochondria within the cells and contributes to the muscle weakness and inflammation accompanying frailty in people living with HIV . This study will examine the impact of six weeks of moderately paced walking on energy production in the cells, inflammation markers and frailty scores in people living with well-controlled HIV who are aged 50 to 65.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 65
* Documentation of HIV infection from Medical Provider
* Currently receiving antiretrovirals
* HIV viral load less than 50 iu/mL for at least six months
* CD4 count at least 350 cell/mm3 for the last six months
* Willing and able to walk at least 30 minutes 3 times weekly within 30 minutes of UMB
* Speaks English

Exclusion Criteria:

* Current smokers
* Weight less than 110 pounds
* Subjects taking long-term corticosteroids equivalent to 10mg/day or more, or immunomodulators
* Subjects with conditions known to affect inflammatory or mitochondrial function other than HIV, such as rheumatoid arthritis, gout, heart failure, chronic obstructive pulmonary disease, chronic kidney disease, diabetes, Parkinson's disease, Alzheimer's disease, active hepatitis, sleep apnea or autoimmune diseases.
* Current drug or alcohol use or dependence or unstable mental health conditions that, in the opinion of the investigator, would interfere with adherence to study requirements

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Mitochondrial Respiration PBMC and platelets | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12
  Change in mitochondrial respiratory capacity after a six-week walking intervention

SECONDARY OUTCOMES:
Inflammation IL-1β | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12 months
  Change in IL-1β after a six-week walking intervention
Inflammation IL-6 | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12
  Change in IL-6 after a six-week walking intervention
Inflammation IL-10 | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12
  Change in IL-10 after a six-week walking intervention
Inflammation TNF-α | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12
  Change in TNF-α after a six-week walking intervention
Inflammation hsCRP | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12
  Change in hsCRP after a six-week walking intervention

OTHER OUTCOMES:
Frailty Related Phenotype | Day 0, Week 6, Week 12 with intervention between weeks 6 and 12
  Change in frailty phenotype score (0-5 with 3 to 5 indicating frailty) after a six-week walking intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Klinedinst, PhD, Principal Investigator — Associate Professor

IPD SHARING:
Plan to Share IPD: No